CLINICAL TRIAL: NCT02963168
Title: A Dose Regimen-Finding Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Activity of Oradoxel Monotherapy in Subjects With Advanced Malignancies
Brief Title: A DRF Study to Evaluate Safety, Tolerability, PK, and Activity of Oradoxel Monotherapy in Subjects w Adv. Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Athenex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KX-ORADOX-003
Record Dates: First submitted 2016-10-07; First posted 2016-11-15 (Estimated); Last update posted 2019-10-17 (Actual); Status verified 2019-01

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oradoxel (Experimental): To determine the MTD of Oradoxel (oral docetaxel and oral HM30181A) when administered once every 3 weeks, then to determine the MTD of Oradoxel (oral docetaxel and oral HM30181A) when administered for two days every three weeks.
  Interventions: Drug: Oradoxel

INTERVENTIONS:
Drug: Oradoxel — oral docetaxel will be supplied in capsules and oral HM30181A-UK tablets
  Other Names: oral docetaxel + oral HM30181A

SUMMARY:
This is a nonrandomized, open-label, dose escalation, safety, activity, and PK study to determine the MTD and optimal dosing regimen of Oradoxel. No control group has been included.

DETAILED DESCRIPTION:
This is a multicenter, open-label, safety, tolerability, pharmacokinetic, and activity study. Eligible subjects will be adults with advanced solid malignancies.

Groups of 3 to 6 subjects will receive a single dose of Oradoxel and will be followed for toxicity. If non linearity in PK is observed, additional subjects will receive Oradoxel as 2 single daily doses once every three weeks. Subjects who tolerate the drug and have stable disease or better response will be eligible to receive ongoing treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. ≥18 years of age
3. Histologically or cytologically confirmed solid tumor that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
4. Docetaxel monotherapy is a reasonable treatment in the judgement of the Investigator
5. Measurable disease as per RECIST v1.1 criteria
6. Able to swallow oral medication as an intact dosage form
7. Adequate hematologic status as demonstrated by not requiring transfusion support or granulocyte-colony stimulating factor (G-CSF) to maintain: Absolute neutrophil count (ANC) ≥1500 cells/mm3, Platelet count ≥100 x 109/L, Hemoglobin (Hgb) ≥10 g/dL
8. Adequate liver function as demonstrated by: Total bilirubin of < upper limit of normal (ULN), Aspartate transaminase (AST) and alanine aminotransferase (ALT) ≤1.5 × ULN, Alkaline phosphatase (ALP) ≤2.5x ULN or <5x ULN if bone metastases are present, Normal serum albumin
9. Adequate renal function as demonstrated by serum creatinine ≤1.5 x ULN or creatinine clearance>60 mL/min as calculated by the Cockroft and Gault formula
10. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
11. Life expectancy of at least 3 months
12. Willing to fast for 6 hours before and 2 hours after Oradoxel administration
13. Females must be postmenopausal (>12 months without menses) or surgically sterile (ie, by hysterectomy and/or bilateral oophorectomy) or, if sexually active, must be using effective contraception (ie, oral contraceptives, intrauterine device, double barrier method of condom and spermicide) and agree to continue use of contraception for 30 days after their last dose of study drug.
14. Sexually active male subjects must use a barrier method of contraception during the study and agree to continue the use of male contraception for at least 30 days after the last dose of study drug.

Exclusion Criteria:

1. Currently taking a prohibited concomitant medication, other than a premedication, that are/is:

   * Strong inhibitors (eg, ketoconazole) or inducers (eg, rifampicin or St. John's Wort) of CYP3A4 (within 2 weeks prior to the start of dosing in the study)
   * Strong P-gp inhibitors or inducers. Subjects who are taking such medications but who are otherwise eligible may be enrolled if they discontinue the medication ≥1 week before dosing and remain off that medication through the end of PK sampling after the administration of the second study treatment
   * An oral medication with a narrow therapeutic index known to be a P-gp substrate within 24 hours prior to start of dosing in the study
2. Unresolved toxicity from prior chemotherapy (subjects must be recovered to ≤ Grade 1 toxicity from previous anticancer treatments or previous investigational products.
3. Planning to receive other medical, surgical, or radiological cancer treatments during the course of this study
4. Received investigational agents within 14 days or 5 half-lives prior to the first study dosing day, whichever is longer
5. Require therapeutic use of anticoagulants
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, clinically significant myocardial infarction within the last 6 months, unstable angina pectoris, clinically significant cardiac arrhythmia, bleeding disorder, chronic pulmonary disease requiring oxygen, or psychiatric illness/social situations that would limit compliance with study requirements
7. Major surgery to the upper gastrointestinal (GI) tract, or have a history of GI disease or other medical condition that, in the opinion of the Investigator, may interfere with oral drug absorption
8. A known history of allergy to docetaxel, Cremophor or polysorbate 80 (Tween 80)
9. Evidence of fluid retention at Screening (including, for example, peripheral edema, pleural effusion, or ascites on physical or radiological examination) or history of severe capillary leak syndrome
10. Any other condition which the Investigator believes would make participation in the study not acceptable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-04-20 (Actual); Primary Completion 2020-03-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD) of Oradoxel based on dose-limiting toxicity (DLT) in subjects with advanced malignancies | 3 weeks
  The MTD will be the highest dose at which no more than 1 of 6 subjects experience a DLT during treatment and Oradoxel pharmacokinetics are acceptable.

SECONDARY OUTCOMES:
Safety assessment using AEs of Oradoxel | Weekly, up to 24 months
Safety assessment using SAEs of Oradoxel | Weekly, up to 24 months
Laboratory evaluation for hematology | Weekly, up to 24 months
Blood chemistry | Weekly, up to 24 months
Urine analysis | Weekly, up to 24 months
Periodic measurements of ECGs | Screening, Day 1, every 6 weeks thereafter up to 24 months
Periodic measurements of vital signs | Weekly, up to 24 months
The incidence of unacceptable toxicity with Oradoxel | 24 months
  Unacceptable toxicity graded according to CTCAE v4.03
The recommended Phase 2 dose (RP2D) of Oradoxel | 24 months
  Upon determination of the overall MTD for Oradoxel, the safety and PK profile of the study treatment from all Treatment Periods will be reviewed to determine the recommended Phase 2 dose.
The amount of docetaxel and HM30181A in blood stream by Area under the plasma concentration versus time curve (AUC) | Part 1: 16 timepoints over 504 hours; Part 2: 26 timepoints over 480 hours
The peak plasma concentration (Cmax) and Minimum plasma concentration (Cmin) | Part 1: 16 timepoints over 504 hours; Part 2: 26 timepoints over 480 hours
A biological half-life or elimination half-life (t1/2) | Part 1: 16 timepoints over 504 hours; Part 2: 26 timepoints over 480 hours
The accumulation ratio (R) | Part 1: 16 timepoints over 504 hours; Part 2: 26 timepoints over 480 hours
The apparent total clearance of the drug from plasma (CL/F) | Part 1: 16 timepoints over 504 hours; Part 2: 26 timepoints over 480 hours
The apparent volume of distribution (Vd/F) | Part 1: 16 timepoints over 504 hours; Part 2: 26 timepoints over 480 hours
To evaluate tumor response | Every 12 weeks, up to 24 months
  Tumor response will be evaluated according to RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: David Cutler, MD, Study Director — Athenex, Inc.
Locations (3):
- United States (3):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic, Rochester, Minnesota
  - Cancer Therapy & Research Center at UTHSCSA, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No